CLINICAL TRIAL: NCT02168738
Title: Bioavailability of DHA-TG (Docosahexaenoic Triglyceride), DHA-PC (Docosahexaenoic Phosphatidylcholine) and AcedoPC (1-acetyl-2-docosahexaenoic-glycerophosphocholine) in Human
Brief Title: Investigation of Docosahexaenoic Acid (DHA) Metabolic Pathway in Human by Using 13C Labeled Molecules
Acronym: AceDoPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012.778
Record Dates: First submitted 2014-03-21; First posted 2014-06-20 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subject
Keywords: nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 13-C labeled PC-DHA (Active Comparator)
  Interventions: Drug: 13-C labeled AceDoPC-DHA; Drug: 13-C labeled TG-DHA; Drug: 13-C labeled PC-DHA
- 13-C labeled TG-DHA (Active Comparator)
  Interventions: Drug: 13-C labeled AceDoPC-DHA; Drug: 13-C labeled TG-DHA; Drug: 13-C labeled PC-DHA
- 13-C labeled AceDoPC-DHA (Experimental)
  Interventions: Drug: 13-C labeled AceDoPC-DHA; Drug: 13-C labeled TG-DHA; Drug: 13-C labeled PC-DHA

INTERVENTIONS:
Drug: 13-C labeled AceDoPC-DHA — Each subject will receive a single dose of either lipid sequentially (according to randomization) a triglyceride (TG-DHA), a phospholipid (PC-DHA) or acetylated lysophosphatidylcholine (AceDoPC) labeled with 13C.
  The dose contains 50 mg 13C-DHA. The wash-out period is four months
Drug: 13-C labeled TG-DHA — Each subject will receive a single dose of either lipid sequentially (according to randomization) a triglyceride (TG-DHA), a phospholipid (PC-DHA) or acetylated lysophosphatidylcholine (AceDoPC) labeled with 13C.
  The dose contains 50 mg 13C-DHA. The wash-out period is four months
Drug: 13-C labeled PC-DHA — Each subject will receive a single dose of either lipid sequentially (according to randomization) a triglyceride (TG-DHA), a phospholipid (PC-DHA) or acetylated lysophosphatidylcholine (AceDoPC) labeled with 13C.
  The dose contains 50 mg 13C-DHA. The wash-out period is four months

SUMMARY:
The purpose of this study is to compare three lipidic forms of DHA in their metabolic pathway in human by using 13C labeled molecules.

The circulating form of DHA plays a major role in his cerebral incorporation. The aim of this research is to confirm that some lipidic forms are best carriers for the cerebral incorporation in studying 13C-DHA distribution in plasma lipids and blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Aged of 60 to 70 years
* Body Mass Index of 20 to 30 kg/m2
* Glycaemic and lipid parameters normal

Exclusion Criteria:

* Smokers more than ten cigarettes/day
* Medical history of personal or family dyslipidemia
* Medication that could interfere with lipid metabolism

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Concentration of 13C-DHA in red blood cells | At Day 1
  6 hours after product ingestion

SECONDARY OUTCOMES:
Concentration of 13C-DHA in plasma lipids | At Day 1
  6 hours after product ingestion
Concentration of 13C-DHA in platelets | At Day 1
  6 hours after product ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes, 165 chemin du Grand Revoyet,, Pierre-Bénite, France

REFERENCES:
- [Result] Hachem M, Nacir H, Picq M, Belkouch M, Bernoud-Hubac N, Windust A, Meiller L, Sauvinet V, Feugier N, Lambert-Porcheron S, Laville M, Lagarde M. Docosahexaenoic Acid (DHA) Bioavailability in Humans after Oral Intake of DHA-Containing Triacylglycerol or the Structured Phospholipid AceDoPC(R). Nutrients. 2020 Jan 18;12(1):251. doi: 10.3390/nu12010251. PMID 31963708
- See also: Related Info — http://www.crnh-rhone-alpes.fr